CLINICAL TRIAL: NCT00893412
Title: Fast-Release Orodispersible Tramadol Tablet (Tradonal Odis®) as Analgesia for Hysterosalpingography : a Randomized, Controlled, Double Blinded Study
Brief Title: Fast-Release Orodispersible Tramadol Tablet (Tradonal Odis®) as Analgesia for Hysterosalpingography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Paul Devroey, UZ Brussel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008/191
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2009-05-06 (Estimated); Status verified 2009-05

CONDITIONS: Infertility; Pain
Keywords: HSG; analgesia; tramadol; metal cannula; balloon catheter
MeSH Terms: conditions — Infertility; Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tramadol + Metal cannula (Active Comparator): Fast-release Orodispersible Tramadol Tablet + Metal cannula
  Interventions: Drug: Fast-release Orodispersible Tramadol Tablet (Tradonal odis®); Procedure: Hysterosalpingography (HSG)
- Placebo + Metal cannula (Placebo Comparator): Placebo + Metal cannula
  Interventions: Procedure: Hysterosalpingography (HSG); Drug: Placebo
- Tramadol + Balloon (Active Comparator): Fast-release Orodispersible Tramadol Tablet + balloon catheter
  Interventions: Drug: Fast-release Orodispersible Tramadol Tablet (Tradonal odis®); Procedure: Hysterosalpingography (HSG)
- Placebo + Balloon (Placebo Comparator): Placebo + balloon catheter
  Interventions: Procedure: Hysterosalpingography (HSG); Drug: Placebo

INTERVENTIONS:
Drug: Fast-release Orodispersible Tramadol Tablet (Tradonal odis®) — 1 tablet of 50 mg Fast-release Orodispersible Tramadol Tablet (Tradonal odis®)
  Other Names: Tradonal odis®
  Arms: Tramadol + Balloon; Tramadol + Metal cannula
Procedure: Hysterosalpingography (HSG) — One HSG using a metal canula or balloon catheter, 30 minutes after tablet
  Other Names: HSG
Drug: Placebo
  Arms: Placebo + Balloon; Placebo + Metal cannula

SUMMARY:
This study evaluates the analgetic effects of the fast-release orodispersible tramadol tablet.

Tramadol acts through a weak affinity for μ receptors and secondly by inhibiting noradrenaline and serotonin neuronal reuptake. It has been used since the 1970s by over 50 million people for the treatment of acute and chronic pain. The orodispersible Tramadol tablet is a new galenic form and is available on the Belgian market for the last three years. Pregastric absorption leads to a quicker onset of action.

So far, evidence shows that pain during and immediately after the Hysterosalpingography (HSG) procedure is only significantly reduced by IV opioid analgesia. This study evaluates the analgetic potential of an orodispersible opioid tablet. This tablet disintegrates rapidly (in around 20-30 seconds) and may be taken without water. Its abuse potential is very low and its respiratory depressant effect is negligible.

DETAILED DESCRIPTION:
Four arm prospective randomized double blinded trial

Patients that need a HSG as part of their diagnostic work-up and are eligible for randomization are counseled about possible participation. After signing the informed consent patients will be randomized in one of the following four groups:

Group 1: Fast-release Orodispersible Tramadol Tablet + metal cannula Group 2: Placebo + metal cannula Group 3: Fast-release Orodispersible Tramadol Tablet + balloon catheter Group 4: Placebo + balloon catheter

Tablets are administered 30 min before the procedure

Primary Endpoint:

* VAS at the six different assessment points

Secondary Endpoint

* adverse effects and complications such as: nausea, vomiting, constipation, drowsiness, respiratory depression, hypotension, allergic reaction and infection

ELIGIBILITY:
Inclusion Criteria:

* > 18 and < 45 years
* Written informed consent

Exclusion Criteria:

* Contra-indication to tramadol, morphine or to other opioids

  * Concomitant use of MAO inhibitors or use less than 2 weeks prior to procedure
  * Use of any other CNS-acting drug
* Contra-indication to radio-contrast medium (allergy)
* Patient already taking analgetics
* History of cervical stenosis
* Presence of pelvic inflammatory disease or any other condition causing pelvic pain
* Clinical and/or laboratory evidence of any major disease
* Pregnant or lactating

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
VAS at the six different assessment points | 24 hours

SECONDARY OUTCOMES:
Adverse effects and complications | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul Devroey, MD, PhD, Study Director — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium